CLINICAL TRIAL: NCT03192397
Title: A Phase Ib/2 Trial of Fludarabine/Melphalan/Total Body Irradiation With Post Transplant Cyclophosphamide as Graft Versus Host Disease Prophylaxis in Matched-Related and Matched-Unrelated Allogeneic Hematopoietic Cell Transplantation
Brief Title: Chemotherapy, Total Body Irradiation, and Post-Transplant Cyclophosphamide in Reducing Rates of Graft Versus Host Disease in Patients With Hematologic Malignancies Undergoing Donor Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 44417; NCI-2017-01069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 44417 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia in Remission; Adult Acute Lymphoblastic Leukemia in Complete Remission; Chronic Myelogenous Leukemia, BCR-ABL1 Positive in Remission; Chronic Myelomonocytic Leukemia in Remission; Graft Versus Host Disease; Hodgkin Lymphoma; Minimal Residual Disease; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Severe Aplastic Anemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Graft vs Host Disease; Hodgkin Disease; Neoplasm, Residual; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Multiple Myeloma; Anemia, Aplastic; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; fludarabine phosphate; Melphalan; Mycophenolic Acid; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (chemotherapy, TBI, cyclophosphamide) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -2 and melphalan hydrochloride IV over 30 minutes on day -2. Patients undergo TBI on day -1.
  STEM CELL INFUSION: Patients undergo allogeneic hematopoietic stem cell transplant on day 0.
  GVHD PROPHYLAXIS REGIMEN: Patients receive cyclophosphamide IV over 2 hours on days 3-4, mycophenolate mofetil IV over 2 hours on days 5-35, and sirolimus IV and then PO once tolerated on days 5-180 with a taper beginning on day 100.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan Hydrochloride; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic stem cell transplant
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan Hydrochloride — Given IV
  Other Names: Alkeran; Alkerana; Evomela
Drug: Mycophenolate Mofetil — Given IV
  Other Names: Cellcept; MMF
Drug: Sirolimus — Given IV and PO
  Other Names: Rapamune
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase Ib/2 trial studies how well chemotherapy, total body irradiation, and post-transplant cyclophosphamide work in reducing rates of graft versus host disease in patients with hematologic malignancies undergoing a donor stem cell transplant. Drugs used in the chemotherapy, such as fludarabine phosphate and melphalan hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft versus host disease). Giving cyclophosphamide after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the cumulative incidence of extensive chronic graft versus host disease (GVHD) at 1 year after transplantation utilizing the novel conditioning/GVHD prophylactic regimen for patients undergoing allogeneic hematopoietic cell transplantation, in patients who do not progress before day 100.

SECONDARY OBJECTIVES:

I. To evaluate clinical response, engraftment rate, progression-free survival (PFS) at one year and, overall survival (OS).

II. To determine the cumulative incidence of relapse. III. To evaluate the day 100 transplant-related mortality rate. IV. To determine the cumulative incidence of grade III-IV acute GVHD.

OUTLINE: This is a dose-escalation study of melphalan hydrochloride.

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -5 to -2 and melphalan hydrochloride IV over 30 minutes on day -2. Patients undergo total body irradiation (TBI) on day -1.

STEM CELL INFUSION: Patients undergo allogeneic hematopoietic stem cell transplant on day 0.

GVHD PROPHYLAXIS REGIMEN: Patients receive cyclophosphamide IV over 2 hours on days 3-4, mycophenolate mofetil IV over 2 hours on days 5-35, and tacrolimus IV and then orally (PO) once tolerated on days 5-180 with a taper beginning on day 100.

After completion of study treatment, patients are followed up for 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a diagnosis of one of the following (one must be yes):

  * Acute myeloid leukemia (AML)
  * Acute lymphoblastic leukemia (ALL)
  * Chronic lymphoblastic leukemia (CLL)
  * Chronic myelogenous leukemia (CML) (chronic phase intolerant or unresponsive to tyrosine kinase inhibitors, accelerated phase, history of blast crisis)
  * Myelodysplastic syndrome (MDS)
  * Non-Hodgkin lymphoma (NHL)
  * Hodgkin lymphoma (HL) (received and failed frontline therapy or failed autologous transplantation or inability to collect enough peripheral blood stem cells [PBSC] for autologous hematopoietic cell transplant [auto-HCT])
  * Multiple myeloma (MM)
  * Severe aplastic anemia
* Histocompatible donor identified:

  * Related donor matched 5/6 or better (A, B, DRB1)
  * Unrelated donor matched 7/8 or better (A, B, C and DRB1)
* Patients with severe aplastic anemia do not have disease requirements; however, if the patient has a mismatched donor, the patient must have had prior therapy with ATG.

The following are eligible for study inclusion:

* Patients with MDS/MPN only require <5% myeloblast on bone marrow evaluation.
* Patients with AML, ALL or CLL may be in CRi, patients with MM may be in VGPR
* Patients with NHL/HL must be in CR

  * Have a Karnofsky performance status score of > 50%
  * Diffusing capacity of the lung for carbon monoxide (DLCO) > 40% predicted, corrected for hemoglobin and/or alveolar ventilation
  * Left ventricular ejection fraction > 40%
  * Bilirubin =< 3 x upper limit of normal
  * Liver alkaline phosphatase =< 3 x upper limit of normal
  * Serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 3 x upper limit of normal
  * Calculated creatinine clearance > 40 cc/min by the modified Cockroft-Gault formula
  * Patient must be cleared pre-transplant by Radiation Oncology to be able to receive 400 cGy
  * Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
  * Patients who have failed a prior autologous or allogeneic transplant are eligible; however, at least 6 months must have elapsed between the start of this reduced intensity conditioning regimen and the last transplant if patient had a prior autologous or myeloablative allogeneic bone marrow transplant (BMT)
  * At least 2 weeks since prior radiation treatment and/or surgery. Appropriate washout of prior chemotherapy per BMT standard of care. If medication is not on the list, go by physician discretion
  * Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Moderate to severe myelofibrosis within 60 days prior to transplant
* Presence of human leukocyte antigen (HLA) antibodies to the donor within 60 days prior to transplant
* Patients who in the opinion of the treating physician are unlikely to comply with the restrictions of allogeneic stem cell transplantation based on formal psychosocial screening. (i.e., serious, uncontrolled psychiatric illness/social situations that would limit compliance with study requirements)
* Uncontrolled diabetes mellitus, cardiovascular disease, active serious infection or other condition which, in the opinion of treating physician, would make this protocol unreasonably hazardous for the patient
* Known human immunodeficiency virus (HIV) positive
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Extensive chronic graft versus host disease (GVHD) | Up to 365 days
  Will be analyzed for each stratum. Will examine in a post-hoc analysis potential chronic GVHD rates of response by human leukocyte antigen (HLA) matching status.

SECONDARY OUTCOMES:
Clinical response assessed as per bone marrow transplant (BMT) standard of care | Up to 4 years
  Will utilize either straight Kaplan-Meier based estimators or extensions of nonparametric survival models to account for competing risks.
Cumulative incidence of grade III-IV acute graft versus host disease (GVHD) | Up to 4 years
  Will be analyzed in a descriptive fashion with means +/- standard deviations or frequency counts. Will examine in a post-hoc analysis potential chronic GVHD rates of response by human leukocyte antigen (HLA) matching status.
Cumulative incidence of relapse | Up to 4 years
  Will be analyzed in a descriptive fashion with means +/- standard deviations or frequency counts.
Engraftment rate assessed as per bone marrow transplant (BMT) standard of care | Up to 4 years
  Will be analyzed in a descriptive fashion with means +/- standard deviations or frequency counts.
Overall survival assessed as per bone marrow transplant (BMT) standard of care | Up to 4 years
  Will utilize either straight Kaplan-Meier based estimators or extensions of nonparametric survival models to account for competing risks.
Progression free survival (PFS) assessed as per bone marrow transplant (BMT) standard of care | At 1 year
  Will utilize either straight Kaplan-Meier based estimators or extensions of nonparametric survival models to account for competing risks.
Treatment-related mortality rates | Up to 4 years
  Will be analyzed in a descriptive fashion with means +/- standard deviations or frequency counts.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Ross, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States